CLINICAL TRIAL: NCT03097588
Title: A Phase II Clinical Trial of NEPA (Netupitant/Palonosetron) for Prevention of Chemotherapy Induced Nausea and Vomiting (CINV) in Patient Receiving the BEAM Conditioning Regimen Prior to Hematopoietic Cell Transplantation (HSCT)
Brief Title: Netupitant and Palonosetron Hydrochloride in Preventing Chemotherapy Induced Nausea and Vomiting in Patients With Cancer Undergoing BEAM Conditioning Regimen Before Stem Cell Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Helsinn Therapeutics (U.S.), Inc (Industry); Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Joseph Bubalo, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00016288; NCI-2017-00548 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00016288 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2017-03-27; First posted 2017-03-31 (Actual); Results first posted 2021-06-03 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-06

CONDITIONS: Malignant Neoplasm
MeSH Terms: conditions — Neoplasms | interventions — netupitant; Palonosetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Supportive care (NEPA) (Experimental): Within 60 minutes before standard of care BEAM treatment, patients receive netupitant and palonosetron hydrochloride PO on days 1, 3, and 6.
  Netupitant: 300 mg, QD, Given PO Palonosetron Hydrochloride: 0.5 mg, QD, Given PO Questionnaire Administration: Ancillary studies
  Interventions: Drug: Netupitant; Drug: Palonosetron Hydrochloride; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Netupitant — 300 mg, Given PO, QD
  Other Names: CID6451149; D05152; RO 67-3189/000
Drug: Palonosetron Hydrochloride — 0.5 mg, Given PO, QD
  Other Names: Aloxi; RS 25259-197
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial studies how well netupitant and palonosetron hydrochloride work in preventing chemotherapy induced nausea and vomiting in patients with cancer undergoing BEAM conditioning regimen before stem cell transplant. Chemotherapy, such as carmustine, cytarabine, etoposide, and melphalan (BEAM), makes people feel sick to their stomach and causes vomiting. Netupitant and palonosetron hydrochloride may reduce the nausea and vomiting caused by the BEAM treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the efficacy of netupitant and palonosetron hydrochloride (NEPA) to prevent nausea and vomiting both during and after a highly emetogenic (BEAM) conditioning regimen for hematopoietic stem cell transplantation (HSCT).

SECONDARY OBJECTIVES:

I. To differentiate response to NEPA over different phases of chemotherapy-induced nausea.

OUTLINE:

Within 60 minutes before standard of care BEAM treatment, patients receive netupitant and palonosetron hydrochloride orally (PO) on days 1, 3, and 6.

After completion of study treatment, patients are followed up at 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be undergoing autologous or allogeneic hematopoietic stem cell transplant (HSCT) with the BEAM conditioning regimen prior to HSCT
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 or Karnofsky Performance Score >= 60%
* Able to swallow oral medications
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Subjects with known hypersensitivity or other allergic reactions attributed to compounds of similar biologic composition to netupitant, palonosetron, dexamethasone, or other agents used in the study
* Subjects who are receiving any other investigational agents or have received another investigational drug in the last 30 days
* Subjects who have had emesis or required antiemetics in the 48 hours prior to starting the BEAM conditioning regimen; patients required to take antipsychotics, appetite stimulants, or other medications with antiemetic effects will also be excluded if those medications cannot be replaced by therapeutic equivalents
* Female subjects who are pregnant, have a positive serum human chorionic gonadotrophin (hCG), or are lactating and intend to breastfeed a child; pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with NEPA
* Human immunodeficiency virus (HIV)-positive subjects on combination antiretroviral therapy are ineligible
* Subjects who have taken a neurokinin antagonist within 14 days prior to beginning the BEAM regimen
* Subjects who have a serum creatinine > 2 x upper limit of normal (ULN)
* Subjects with severe renal failure or end stage renal disease (estimated GFR [glomerular filtration rate] of < 30 mL/min) as estimated by the Cockcroft-Gault formula
* Subjects with severe hepatic insufficiency (Child Pugh score > 9)
* Subjects who have been reported > 5 alcoholic drinks daily for the last year
* Subjects who have concurrent illness requiring systemic corticosteroid use other than the planned dexamethasone during conditioning therapy
* Subjects with gastrointestinal conditions that might result in malabsorption of the study drug
* Subjects with a history of anxiety-induced ("anticipatory") nausea and vomiting
* Subjects on strong CYP 3A4 inducers or inhibitors who are unable to have those agents replaced with clinical alternatives prior to beginning the study; length of washout period will be 7 days; notably, in the case of allogeneic transplant recipients requiring cyclosporine or tacrolimus, no empiric dose adjustments will be required due to close level monitoring and adjustments, that are standard in Oregon Health & Science University (OHSU) protocols
* Subjects unable to discontinue benzodiazepines as antiemetics will not be allowed; additional antiemetics will be allowed for rescue but not for prophylaxis
* Subjects with personal or family history of QT prolongation, uncorrected electrolyte abnormalities, congestive heart failure, bradyarrhythmia, conduction disturbances and those taking antiarrhythmic medicinal products or other medicinal products that lead to QT prolongation or electrolyte abnormalities; relevant information will be collected as part of subject medical history

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2017-04-27 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-03-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Bubalo, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Supportive Care (NEPA)
Started | 43
Completed | 42
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Supportive Care (NEPA)
Number analyzed (Participants) | 43
Age, Continuous [Mean (Full Range); unit: years] | 55 [23 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 27
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 41
  Race: Black or African American | 1
  Race: Native Hawaiian/other Pacific Highlander | 1

OUTCOME MEASURES:

1. Primary Outcome: Complete Response (CR) Defined as no Emesis and no Rescue Therapy
Description: Number of subjects that reached a complete response (CR), defined as having no emesis and no rescue therapy.
Time Frame: Up to 5 days post chemotherapy
Measure: Count of Participants; unit: Participants
Arm/Group | Supportive Care (NEPA)
Number analyzed (Participants) | 42
Participants | 13

2. Secondary Outcome: CR (Acute Phase)
Description: Number of subjects that reached a complete response (CR), defined as having no emesis and no rescue therapy from 0 to 144 hours (acute phase) of the study drug administration.
Time Frame: Up to 144 hours post-study drug administration on day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Supportive Care (NEPA)
Number analyzed (Participants) | 42
Participants | 12

3. Secondary Outcome: CR (Delayed Phase)
Description: Number of subjects that reached a complete response (CR), defined as having no emesis and no rescue therapy from 145 hours up to 264 hours (delayed phase) of the study drug administration.
Time Frame: From 145 hours up to 264 hours post-study drug administration on day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Supportive Care (NEPA)
Number analyzed (Participants) | 42
Participants | 1

4. Secondary Outcome: Complete Protection (CP) Rate Defined as CR Plus no Nausea
Description: Number of subjects that reached a complete response (CR), defined as having no emesis and no rescue therapy from 0 to 264 hours of the study drug administration.
Time Frame: Up to 264 hours post-study drug administration on day 1
Population: 42 participants completed the study and therefore were analyzed for response.
Measure: Count of Participants; unit: Participants
Arm/Group | Supportive Care (NEPA)
Number analyzed (Participants) | 42
Participants | 3

5. Other Pre Specified Outcome: Number of Participants With Emetic Episodes and Received Rescue Agents
Description: The number of participants that had emetic episodes and received rescue agents (medications).
Time Frame: Up to 264 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Supportive Care (NEPA)
Number analyzed (Participants) | 43
Participants
  Number of participants who had emetic episodes | 8
  Number of participants who were given rescue meds | 36

6. Other Pre Specified Outcome: Number of Participants With Emetic Episodes and Received Rescue Agents (Acute Phase)
Description: The number of participants that had emetic episodes and received rescue agents (medications) (acute phase: for 0 to 144 hours timeframe of study drug administration)
Time Frame: Up to 144 hours post-study drug administration on day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Supportive Care (NEPA)
Number analyzed (Participants) | 43
Participants
  Number of participants who had an emetic episode in acute phase | 0
  Number of participants who were given rescue meds in acute phase | 13

7. Other Pre Specified Outcome: Number of Participants With Emetic Episodes and Received Rescue Agents (Acute Phase)
Description: The number of participants that had emetic episodes and received rescue agents (medications) (for 0 to 24 hours timeframe of study drug administration)
Time Frame: Up to 24 hours post-study drug administration on day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Supportive Care (NEPA)
Number analyzed (Participants) | 43
Participants
  Number of participants that had emetic episodes | 0
  Number of participants that were given rescue meds- | 2

8. Other Pre Specified Outcome: Number of Participants With Emetic Episodes and Received Rescue Agents (Delayed Phase)
Description: The number of participants that had emetic episodes and received rescue agents (medications) during the delayed phase (for 145 hours up to 264 hours timeframe)
Time Frame: From 145 hours up to 264 hours post-study drug administration on day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Supportive Care (NEPA)
Number analyzed (Participants) | 43
Participants
  The number of participants that had an emetic episode | 8
  The number of participants that were given rescue meds | 23

9. Other Pre Specified Outcome: Mean Levels of Nausea Per Day Assessed by Chemotherapy Induced Nausea and Vomiting Questionnaire
Description: The mean level of nausea per day assessed by chemotherapy induced nausea and vomiting questionnaire. The full range of nausea level score on the questionnaire was from minimum value of 0 to a maximum value of 10. 0= no nausea or vomiting, and 10= worst nausea and vomiting. Higher score means a worse outcome.
Time Frame: Up to 11 days
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Supportive Care (NEPA)
Number analyzed (Participants) | 43
score on a scale | 2.79 [0 to 10]

10. Other Pre Specified Outcome: Time to First Emesis and Time to Receiving First Rescue Medication
Description: Will be depicted via Kaplan-Meier curves showing the percentage of patients who had no emesis or rescue medication use for the acute and delayed time periods.
Time Frame: Up to 264 hours
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | Supportive Care (NEPA)
Number analyzed (Participants) | 43
Hours
  Median time to receiving rescue medication | 148.4 [130.2 to 185.1]
  Time to first emesis | 216 [168 to 240]

11. Other Pre Specified Outcome: Time to Receiving First Rescue Medication and First Emesis
Description: as for outcome 10
Time Frame: Up to 264 hours
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Supportive Care (NEPA)
Number analyzed (Participants) | 43
Hours
  Mean time to first rescue medication | 143 (55.27)
  Mean time to first emesis | 8.9 (0.83)

ADVERSE EVENTS:
Time Frame: Adverse event collection will begin when subject takes their first dose of study drug and continues until the subject completes the End of Study visit, up to 20 days, or until 1 month if toxicity on trial occurs, whichever comes later. Maximum duration up to 1 month.
Arm/Group | Supportive Care (NEPA)
All-Cause Mortality (participants affected / at risk) | 1/43
Serious Adverse Events (participants affected / at risk) | 1/43
Other Adverse Events (participants affected / at risk) | 43/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Supportive Care (NEPA) (N=43)
Vomiting (Gastrointestinal disorders) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Transfusion Related Acute Lung Injury (Investigations) | 1 (1)
Pulseless Electrical Activity (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Supportive Care (NEPA) (N=43)
Abdominal cramping (Gastrointestinal disorders) | 6 (6)
Colitis (Gastrointestinal disorders) | 18 (18)
Anemia (Blood and lymphatic system disorders) | 35 (35)
CD4 Lymphocytes decreased (Blood and lymphatic system disorders) | 6 (6)
Febrile Neutropenia (Blood and lymphatic system disorders) | 12 (12)
Lymphocyte count reduced (Blood and lymphatic system disorders) | 32 (32)
Neutropenia (Blood and lymphatic system disorders) | 33 (33)
Leukopenia (Blood and lymphatic system disorders) | 41 (41)
Hypertension (Cardiac disorders) | 3 (3)
Fatigue (General disorders) | 4 (4)
Bacteremia (Infections and infestations) | 5 (5)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 6 (6)
Hypokalemia (Metabolism and nutrition disorders) | 6 (6)
Hypophosphatemia (Metabolism and nutrition disorders) | 6 (6)
Thrombocytopenia (Blood and lymphatic system disorders) | 39 (39)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-27): https://cdn.clinicaltrials.gov/large-docs/88/NCT03097588/Prot_SAP_000.pdf